CLINICAL TRIAL: NCT02685085
Title: Combined Method for Induction of Labor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Woman's Health University Hospital, Egypt (Other)
Responsible Party: Principal Investigator, Dina Mohamed Refaat Dakhly, Lecturer of Obstetrics and Gynecology, Woman's Health University Hospital, Egypt
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FM0702116
Record Dates: First submitted 2016-02-09; First posted 2016-02-18 (Estimated); Last update posted 2016-02-18 (Estimated); Status verified 2016-02

CONDITIONS: Induced Labor
MeSH Terms: interventions — Misoprostol; Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Misoprostol (Experimental): in this group misoprostol 25 ug will be administrated for induction of labor every 6 hours
  Interventions: Drug: Misoprostol ( Prostaglandin E2)
- Foley's catheter (Experimental): In this group foley's catheter 30 cc will be used for induction of labor
  Interventions: Device: Foley's catheter
- Combined (Experimental): Both misoprostol 25 ug and foley's catheter will be used for induction
  Interventions: Drug: Misoprostol ( Prostaglandin E2); Device: Foley's catheter

INTERVENTIONS:
Drug: Misoprostol ( Prostaglandin E2)
  Other Names: Cytotec
  Arms: Combined; Misoprostol
Device: Foley's catheter
  Arms: Combined; Foley's catheter

SUMMARY:
Induction of labor is performed via the vaginal misorostol 25 ug/ 6 hours and intracervical foley's cather administration and both techniques performed together.

ELIGIBILITY:
Inclusion Criteria:

* females presenting for induction of labor

Exclusion Criteria:

* previous cesarean section
* previous uterine scars e.g. myomectomy
* refusal to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Duration of induction of labor | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dina MR Dakhly, MD, Principal Investigator — Cairo University
Locations (1):
- Kasr el aini hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided